CLINICAL TRIAL: NCT06874946
Title: A Phase I Dose-Escalation and Phase II Study of Nanobody-Based CD5-Targeted CAR-T Cells for the Treatment of Relapsed or Refractory T-Cell Acute Lymphoblastic Leukemia/Lymphoma (T-ALL/LBL) - The CONQUER Trial
Brief Title: Nanobody-Based Anti-CD5 CAR-T for Relapsed/Refractory T-ALL/LBL
Acronym: Phase I/II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiangyu Zhao, Deputy Hospital Director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHD001-001
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Precursor T-Cell Lymphoblastic Leukemia-Lymphoma
Keywords: R/R T-ALL/LBL; CD5
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: anti CD5 CAR-T cells, eligible patients will be treated with CD5-targeted CAR-T cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD5-targeted CAR-T cells (Experimental): Eligible patients will receive a single infusion of CD5-targeted CAR-T cells at 3+3 dose-escalation design.
  Phase II: Patients will receive CD5-targeted CAR-T cells at the RP2D.
  Interventions: Biological: CD5-targeted CAR-T cells

INTERVENTIONS:
Biological: CD5-targeted CAR-T cells — Phase I: Eligible patients will receive a single infusion of CD5-targeted CAR-T cells at one of three dose levels (0.5 × 10⁶ cells/kg, 1.0 × 10⁶ cells/kg, or 2.0 × 10⁶ cells/kg) following fludarabine and cyclophosphamide (FC) lymphodepleting chemotherapy. A 3+3 dose-escalation design will be used to determine the recommended Phase II dose (RP2D) based on safety, dose-limiting toxicities (DLTs), and preliminary efficacy.
  Phase II: Patients will receive CD5-targeted CAR-T cells at the RP2D following FC lymphodepleting chemotherapy.

SUMMARY:
To observe the safety and efficacy of Nanobody-Based CD5-targeted chimeric antigen receptor T cells in the treatment of refractory or relapsed T-ALL/LBL.

DETAILED DESCRIPTION:
This Phase I/II study aims to evaluate the safety, tolerability, and efficacy of Nanobody-Based CD5 Chimeric Antigen Receptor (CAR) T-cell therapy in patients with relapsed or refractory (R/R) T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL).

In the Phase I portion, a 3+3 dose-escalation design will be utilized to assess the safety profile and determine the optimal dose of Nanobody-Based CD5 CAR-T cells. The recommended Phase II dose (RP2D) will be established based on safety data, dose-limiting toxicities (DLTs), and preliminary efficacy outcomes.

The Phase II portion will then evaluate the efficacy of Nanobody-Based CD5 CAR-T therapy at the RP2D. The primary and secondary endpoints will include:

Overall response rate (ORR) Disease-free survival (DFS) Overall survival (OS) Comprehensive safety assessments will be conducted throughout the study, with a particular focus on cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS).

By investigating Nanobody-Based CD5 CAR-T therapy, this study aims to address the significant unmet clinical need for effective treatment options in patients with R/R T-ALL/LBL and provide insights into its potential as a novel immunotherapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or guardian understands and voluntarily signs the informed consent form (ICF).
2. Male or female, aged 3-70 years at the time of signing the ICF (inclusive).
3. Expected survival of at least 12 weeks.
4. ECOG performance status of 0-2 at the time of ICF signing.
5. Diagnosis of relapsed/refractory T-cell lymphoblastic leukemia/lymphoma (R/R T-ALL/LBL) confirmed at screening and meeting at least one of the following criteria:

   1. Bone marrow involvement: Morphologic examination shows ≥5% lymphoblasts, and/or
   2. Cerebrospinal fluid (CSF) involvement: Tumor cells detected in CSF, and/or
   3. Extramedullary disease: Presence of measurable lesions (lymph node/mass ≥1.5 cm in axial diameter or extranodal lesion ≥1 cm in axial diameter).
   4. CD5 expression: Tumor cells in bone marrow, peripheral blood, or CSF are CD5-positive by flow cytometry, and/or lymph node/mass or extranodal lesions are CD5-positive by pathology.
6. Adequate major organ function, defined as:

   1. AST and ALT ≤5× upper limit of normal (ULN).
   2. Total bilirubin ≤2× ULN.
   3. Renal function: Serum creatinine clearance ≥60 mL/min (Cockcroft-Gault formula) or creatinine ≤1.5× ULN.
7. Blood oxygen saturation >92%.
8. Reproductive health requirements:

   * Fertile men and women of childbearing potential must agree to use effective contraception from ICF signing until 2 years after study drug administration.
   * Women of childbearing potential (pre-menopausal or within 2 years post-menopause) must have a negative blood pregnancy test at screening.

Exclusion Criteria:

1. History of central nervous system (CNS) diseases, including but not limited to:

   * Epilepsy
   * Paralysis
   * Aphasia
   * Stroke
   * Severe brain injury
   * Dementia
   * Parkinson's disease
   * Neuropathy
2. History of autoimmune diseases requiring systemic immunosuppressive therapy within 2 years prior to signing the ICF, including but not limited to:

   * Crohn's disease
   * Rheumatoid arthritis
   * Systemic lupus erythematosus (SLE)
   * Systemic sclerosis
   * Inflammatory bowel disease (IBD)
   * Vasculitis
   * Psoriasis
3. Presence of any uncontrolled active infection at the time of signing the ICF or within 4 weeks prior to apheresis that requires antibiotic, antiviral, or antifungal treatment.
4. Positive virological or infectious disease markers, including:

   * Hepatitis B virus (HBV): Subjects with positive HBsAg or HBcAb-positive at screening must have undetectable HBV DNA in peripheral blood to be eligible; otherwise, they should be excluded.
   * Hepatitis C virus (HCV): Subjects with positive HCV antibodies and detectable HCV RNA should be excluded.
   * Human immunodeficiency virus (HIV) antibody-positive subjects should be excluded.
   * Cytomegalovirus (CMV) DNA test-positive subjects should be excluded.
   * Epstein-Barr virus (EBV) DNA test-positive subjects should be excluded.
   * Positive serological or non-specific antibodies for Treponema pallidum (syphilis).
5. Clinically significant cardiovascular diseases, including any of the following:

   1. QTc interval ≥480 ms (Fridericia correction formula)
   2. New York Heart Association (NYHA) Class II or higher heart failure
   3. Unstable angina or acute myocardial infarction within 6 months prior to signing the ICF
   4. Left ventricular ejection fraction (LVEF) <50%
   5. Poorly controlled hypertension (as determined by the investigator)
   6. Clinically significant arrhythmias or those requiring antiarrhythmic treatment, including:

      * Persistent ventricular tachycardia
      * Ventricular fibrillation
      * Torsades de pointes
      * Complete left bundle branch block
6. History of severe hypersensitivity or allergy to any components of the study drug.
7. Receipt of any investigational drug therapy or other systemic antitumor therapy within 4 weeks before apheresis (or 5 half-lives of the drug, whichever is longer, as determined by the investigator).
8. Receipt of extensive radiotherapy within 4 weeks prior to signing the ICF, except for palliative radiotherapy for non-target lesions within 2 weeks before signing the ICF or as expected during the study.
9. Unresolved toxicity from prior antitumor therapy that has not returned to Grade 1 or baseline levels at the time of signing the ICF, except for hair loss and pigmentation (per NCI-CTCAE v5.0).
10. Requirement for systemic corticosteroids or other immunosuppressive therapy (≥10 mg/day prednisone or equivalent) within 3 days prior to apheresis or during the study period, except for:

    1. Intranasal, inhaled, or topical steroids, or localized steroid injections (e.g., intra-articular injections)
    2. Systemic corticosteroids ≤10 mg/day prednisone (or equivalent physiological dose)
    3. Steroids as prophylaxis for allergic reactions (e.g., pre-medication before contrast-enhanced CT)
    4. Steroids used for symptomatic treatment of transfusion-related reactions
11. Major surgery within 4 weeks prior to signing the ICF (excluding routine biopsy procedures) or planned major surgery during the study period.
12. History of active tuberculosis infection within 1 year prior to signing the ICF, except for subjects with a history of tuberculosis more than 1 year ago, provided that the investigator determines there is no evidence of active tuberculosis.
13. History of other primary malignancies within 5 years prior to signing the ICF, except for:

    1. Adequately treated carcinoma in situ of the cervix
    2. Localized basal cell carcinoma or squamous cell carcinoma of the skin
14. Receipt of live-attenuated or inactivated vaccines within 4 weeks before signing the ICF or planned vaccination during the screening period.
15. Any other condition or complication that, in the investigator's judgment, may affect adherence to the study protocol or make the subject unsuitable for participation.
16. Pregnancy or lactation.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT (Dose-Limiting Toxicity) | Day28 after CAR-T cell infusion
  CRS and ICANS will be assessed per ASTCT (2019), while other AEs follow CTCAE v5.0. DLTs are CAR-T-related AEs that occur within 28 days post-infusion and meet the following criteria:
  Grade 4+ CRS, or Grade 3 CRS unresolved to ≤ Grade 2 within 7 days. Grade 3+ non-hematologic toxicity unresolved to ≤ Grade 2 within 7 days. Grade 4+ ICANS, or Grade 3 ICANS unresolved to ≤ Grade 2 within 3 days. Grade 3+ hypersensitivity reaction. Any unexpected toxicity requiring study discontinuation.
  Exemptions:
  Rapid hypersensitivity resolving to ≤ Grade 2 in 2 hours. Reversible Grade 3 AEs lasting ≤7 days. Transient CRS-related organ dysfunction, resolving in ≤7 days per SRC.
  All DLTs are reviewed by the Safety Review Committee (SRC).
Overall Response Rate (ORR) | Within 3 months after CAR-T cell infusion
  ORR is defined as the proportion of patients achieving Complete Remission (CR), Complete Remission with Incomplete Hematologic Recovery (CRi), or Morphologic Leukemia-Free State (MLFS) per European LeukemiaNet (ELN) 2022 for T-ALL and Lugano/Lyric 2016 for T-LBL.
  CR: <5% blasts in bone marrow, no circulating blasts/extramedullary disease, ANC >1.0 × 10⁹/L, platelets >100 × 10⁹/L, MRD-negative.
  CRi: Meets CR but lacks full hematologic recovery. MLFS: <5% blasts, no hematologic recovery required. Lugano 2016 (T-LBL): CR = complete metabolic response on PET-CT; PR = ≥50% tumor reduction.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Within 2-year after CAR-T cell infusion
  Progression-Free Survival (PFS) is defined as the time from the date of first documented Complete Remission (CR), Complete Remission with Incomplete Hematologic Recovery (CRi), or Morphologic Leukemia-Free State (MLFS) until the date of bone marrow (BM) or peripheral blood (PB) relapse, extramedullary disease (EMD) progression, or death from any cause, whichever occurs first.
  PFS will be assessed according to European LeukemiaNet (ELN) 2022 criteria for T-ALL and Lugano/Lyric 2016 criteria for T-LBL.
Overall Survival (OS) | Within 2-year after CAR-T cell infusion
  Overall Survival (OS) is defined as the time from the date of CD5-targeted CAR-T cell infusion until death from any cause. Patients alive at the time of analysis will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No